CLINICAL TRIAL: NCT04672668
Title: Correlation Between the Volume Flow of the CFA After Angioplasty of Critical Ischemic Limb and Wound Healing
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Chen Speter, dr, Sheba Medical Center
Other Study IDs: SHEBA-20-7318-CP-CTIL
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Wound Heal, Duplex Volume Flow
MeSH Terms: interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: duplex ultrasound for the common femoral artery — duplex ultrasound for the common femoral artery before and after the angiography

SUMMARY:
in our study we are examining the volume flow of the common femoral artery before and after angigraphy of a critical ischemic limb, as a predictor for wound healing after the treatment

DETAILED DESCRIPTION:
All patients with threatened limbs, that was decided upon to have angioplasty will be asked to sign consent form to participate in this study.

Before having the angioplasty, all participants will be examined with ultrasound duplex to determent their common femoral artery volume flow. Day after the angioplasty, they will be reexamined (this is the usual practice) to detriment the new volume flow in the CFA.

The participents examinations in the outpatient clinics will be documented and time for healing will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients with threatened limbs, that was decided upon to have angioplasty .

Exclusion Criteria:

* those who are not willing to sign a consent form to participate in this study

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with threatened limbs, having angioplasty .
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
wound healing | 12 months
  physical examination

CONTACTS AND LOCATIONS:
Overall Officials: moshe halak, dr, Study Chair — sheba health center
Locations (1):
- Sheba Health Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No